CLINICAL TRIAL: NCT00989989
Title: A Randomized, Double-masked, Multicenter, Laser Controlled Phase III Study Assessing the Efficacy and Safety of Ranibizumab (Intravitreal Injections) as Adjunctive and Monotherapy in Patients With Visual Impairment Due to Diabetic Macular Edema
Brief Title: Efficacy and Safety of Ranibizumab (Intravitreal Injections) in Patients With Visual Impairment Due to Diabetic Macular Edema
Acronym: REVEAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002D2303
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-09

CONDITIONS: Diabetic Macular Edema
Keywords: DME; Diabetic; macula; edema; ranibizumab; REVEAL
MeSH Terms: conditions — Edema | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Adjunctive treatment (Experimental): Adjunctive administration of ranibizumab 0.5 mg intravitreal injections and active laser.
  Interventions: Drug: Ranibizumab; Procedure: Laser photocoagulation
- Monotherapy treatment (Experimental): Monotherapy ranibizumab 0.5 mg intravitreal injections plus sham laser.
  Interventions: Drug: Ranibizumab; Procedure: Sham laser photocoagulation
- Laser control (Active Comparator): Active laser treatment plus sham intravitreal injections.
  Interventions: Procedure: Laser photocoagulation; Drug: Sham ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab 0.5 mg intravitreal injection at day 1, month 1 and month 2. If stable vision not reached at month 3, one injection per month continued until stable vision was reached. Intravitreal injections re-initiated if needed.
  Arms: Adjunctive treatment; Monotherapy treatment
Procedure: Laser photocoagulation — Active laser treatment administered at day 1. Subsequent laser treatments administered if needed at intervals no shorter than 3 months from previous laser treatment.
  Arms: Adjunctive treatment; Laser control
Drug: Sham ranibizumab — Sham intravitreal injections to ranibizumab at day 1, month 1 and month 2. Intravitreal injections re-initiated if needed.
  Arms: Laser control
Procedure: Sham laser photocoagulation — Sham laser treatment administered at day 1.
  Arms: Monotherapy treatment

SUMMARY:
This study was designed to confirm the efficacy and safety of ranibizumab (0.5 mg) as adjunctive therapy when added to laser photocoagulation and/or as monotherapy in Asian patients with visual impairment due to Diabetic Macular Edema (DME).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or Type 2 diabetes mellitus according to American Diabetes Association (ADA) or World Health Organization (WHO) guidelines with HbA1c not more than 10.0% at screening (Visit 1). Patients should be on diet, exercise, and/or pharmacological treatment for diabetes.
* Patients with visual impairment due to focal or diffuse Diabetic Macular Edema in at least one eye who are eligible for laser treatment in the opinion of the investigator. If both eyes are eligible, the one with the worse visual acuity, as assessed at Visit 1, will be selected for study treatment unless, based on medical reasons, the investigator deems the other eye the more appropriate candidate for study treatment.
* The study eye must fulfill the following criteria at Visit 1:

  * Best-Corrected Visual Acuity (BCVA) score between 78 and 39 letters, inclusively, using Early Treatment of Diabetic Retinopathy (ETDRS) chart-like visual acuity testing charts at a testing distance of 4 meters (approximate Snellen equivalent of 20/32 to 20/160).
  * Decrease in vision is due to DME and not due to other causes, in the opinion of the investigator.
  * Medication for the management of diabetes must have been stable within 3 months prior to randomization and is expected to remain stable during the course of the study.

Exclusion Criteria:

* Ocular concomitant conditions/ diseases:

  * Concomitant conditions in the study eye which could, in the opinion of the investigator, prevent the improvement of visual acuity on study treatment.
  * Active intraocular inflammation in either eye.
  * Any active infection in either eye.
  * History of uveitis in either eye.
  * Uncontrolled glaucoma in either eye.
* Ocular treatments:

  * Panretinal laser photocoagulation in the study eye within 6 months prior to or during the study.
  * Focal/grid laser photocoagulation in the study eye within 3 months prior to study entry.
* Systemic conditions or treatments:

  * History of stroke
  * Renal failure requiring dialysis or renal transplant or renal insufficiency with creatinine level > 2.0 mg/dL.
  * Untreated diabetes mellitus
  * Blood pressure systolic > 160 mmHg or diastolic > 100 mmHg
* Compliance/ Administrative:

  * Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis
Locations (35):
- China (9):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Changsha
  - Novartis Investigative Site, Chengdu
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Hangzhou
  - Novartis Investigational Site, Shanghai
  - Novartis Investigative Site, Wenzhou
  - Novartis Investigative Site, Xi'an
- Novartis Investigative Site, Hong Kong, Hong Kong
- Japan (20):
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Chiyoda-ku
  - Novartis Investigative Site, Chūōku
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Fukushima
  - Novartis Investigative Site, Hirakata
  - Novartis Investigative Site, Kita-gun
  - Novartis Investigative Site, Kobe
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Mitaka
  - Novartis Investigative Site, Nagoya
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Ōtsu
  - Novartis Investigative Site, Shimotsuke
  - Novartis Investigative Site, Shinjuku-ku
  - Novartis Investigative Site, Suita
  - Novartis Investigative Site, Toyko
  - Novartis Investigative Site, Urayasu
  - Novartis Investigative Site, Wakayama
  - Novartis Investigative Site, Yamagata
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative Site, Taipei

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Started | 132 | 133 | 131
Completed | 114 | 123 | 108
Not Completed | 18 | 10 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control | Total
Number analyzed (Participants) | 132 | 133 | 131 | 396
Age Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.52) | 60.7 (9.37) | 61.5 (9.68) | 61.1 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 52 | 56 | 173
  Male | 67 | 81 | 75 | 223

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline of Best-Corrected Visual Acuity (BCVA) Over 12 Months (From Month 1 to Month 12 Compared to Baseline)
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A positive average change from baseline of BCVA indicates improvement.
Time Frame: 12 months
Population: The Full Analysis Set (FAS) consisted of all randomized patients who received at least one application of study treatment (ranibizumab or sham injection and/or laser or sham treatment) and had at least one post-baseline assessment for Best-Corrected Visual Acuity.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Number analyzed (Participants) | 129 | 133 | 128
Letters | 5.7 (7.20) | 5.9 (6.02) | 1.4 (6.49)

2. Secondary Outcome: Change From Baseline on Central Retinal Subfield Thickness (CRST) at Month 12
Description: Central Retinal Subfield Thickness (CRST) was measured using Optical Coherence Tomography (OCT) in micrometers. A negative change from baseline of CRST indicates improvement.
Time Frame: 12 months
Population: The Full Analysis Set consisted of all randomized patients who received at least one application of study treatment (ranibizumab or sham injection and/or laser or sham treatment) and had Central Retinal Subfield Thickness value with signal strength ≥ 5 for Carl Zeiss Optical Coherence Tomography 3 system.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Number analyzed (Participants) | 115 | 116 | 115
micrometers | -171.8 (160.85) | -134.6 (131.17) | -57.2 (118.60)

3. Secondary Outcome: Percent of Participants With Anatomical Changes in Intra-retinal Cysts at End of Study Compared to Baseline
Description: Presence or absence of intra-retinal cysts in any of the 6 sections of the study eye was measured using Optical Coherence Tomography (OCT). A complete resolution or decrease from baseline of intra-retinal cysts indicates improvement.
Time Frame: Up to 12 months
Population: The Full Analysis Set consisted of all randomized patients who received at least one application of study treatment (ranibizumab or sham injection and/or laser or sham treatment) and had intra-retinal cysts in any of the 6 sections of the study eye at baseline - not applicable means there was no intra-retinal cyst at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Number analyzed (Participants) | 78 | 77 | 77
percentage of participants
  complete resolution | 19.5 | 21.8 | 6.5
  decrease | 40.3 | 42.3 | 35.1
  no change | 5.2 | 5.1 | 15.6
  increase | 1.3 | 1.3 | 10.4
  not applicable | 2.6 | 1.3 | 0
  missing | 31.2 | 28.2 | 32.5

4. Secondary Outcome: Percent of Participants With Anatomical Changes in Sub-retinal Fluid at End of Study Compared to Baseline
Description: Presence or absence of sub-retinal fluid in any of the 6 sections of the study eye was measured using Optical Coherence Tomography (OCT). A complete resolution or decrease from baseline of sub-retinal fluid indicates improvement.
Time Frame: Up to 12 months
Population: The Full Analysis Set consisted of all randomized patients who received at least one application of study treatment (ranibizumab or sham injection and/or laser or sham treatment) and had sub-retinal fluid in any of the 6 sections of the study eye at baseline. Not applicable means there was no sub-retinal fluid at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Number analyzed (Participants) | 22 | 27 | 16
percentage of participants
  complete resolution | 13.6 | 33.3 | 25.0
  decrease | 18.2 | 11.1 | 18.8
  no change | 4.5 | 0 | 6.3
  increase | 0 | 0 | 0
  not applicable | 31.8 | 18.5 | 12.5
  missing | 31.8 | 37.0 | 37.5

5. Secondary Outcome: Percent of Participants With Visual Acuity Above 73 Letters at Month 12
Description: Best Corrected Visual Acuity (BCVA) was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like chart at baseline and month 12 while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. BCVA above 73 letters at month 12 indicates a positive outcome.
Time Frame: 12 months
Population: The Full Analysis Set consisted of all randomized patients who received at least one application of study treatment (ranibizumab or sham injection and/or laser or sham treatment)and had at least one post-baseline assessment for Best-Corrected Visual Acuity.
Measure: Number; unit: percentage of participants
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Number analyzed (Participants) | 122 | 121 | 118
percentage of participants | 20.5 | 16.5 | 8.5

6. Secondary Outcome: Percent of Participants Who Gained >= 10 Letters at Month 12 Compared to Baseline
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A gain of 10 or more BCVA letters from baseline indicates improvement. A BCVA of 84 letters or more at Month 12 indicates improvement.
Time Frame: 12 months
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Number analyzed (Participants) | 129 | 133 | 128
Percentage of participants | 37.2 (37.2) | 33.8 (33.8) | 13.3 (13.3)

7. Secondary Outcome: Percent of Participants Who Lost >= 10 Letters at Month 12 Compared to Baseline
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A loss of 10 or more BCVA letters from baseline indicates worsening.
Time Frame: 12 months
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Number analyzed (Participants) | 129 | 133 | 128
Percentage of participants | 5.4 | 3.0 | 6.3

8. Secondary Outcome: Percent of Participants Who Gained >= 15 Letters at Month 12 Compared to Baseline
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A gain of 15 or more BCVA letters from baseline indicates improvement. A BCVA of 84 letters or more at Month 12 indicates improvement.
Time Frame: 12 months
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Number analyzed (Participants) | 129 | 133 | 128
Percentage of participants | 17.8 | 18.8 | 7.8

9. Secondary Outcome: Percent of Participants Who Lost >= 15 Letters at Month 12 Compared to Baseline
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A loss of 15 or more BCVA letters from baseline indicates worsening.
Time Frame: 12 months
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Number analyzed (Participants) | 129 | 133 | 128
Percentage of participants | 3.9 | 1.5 | 3.9

10. Secondary Outcome: Best-Corrected Visual Acuity (BCVA) Mean Change From Baseline at Month 12
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement.
Time Frame: 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Number analyzed (Participants) | 129 | 133 | 128
Letters | 6.4 (10.67) | 6.6 (7.68) | 1.8 (8.27)

11. Secondary Outcome: Patient Outcome Measure Euro Quality of Life Questionnaire (EQ-5D)
Description: The Euro Quality of Life Questionnaire (EQ-5D) standardized instrument was utilized to measure health outcomes related to mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Participants self-rate their health on a visual, vertical analogue scale from 0 to 100 where the endpoints are labeled "Best imaginable health state" (100) and "worst imaginable health state" (0).
Time Frame: 12 months
Population: The Full Analysis Set consisted of all randomized patients who received at least one application of study treatment (ranibizumab or sham injection and/or laser or sham treatment) and had at least one post-baseline assessment for Best-Corrected Visual Acuity.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adjunctive Treatment | Monotherapy Treatment | Laser Control
Number analyzed (Participants) | 127 | 129 | 125
units on a scale | 2.8 (14.38) | -1.1 (12.74) | 1.0 (13.90)

ADVERSE EVENTS:
Arm/Group | Monotherapy Treatment | Adjunctive Treatment | Laser Control
Serious Adverse Events (participants affected / at risk) | 21/133 | 22/132 | 19/128
Other Adverse Events (participants affected / at risk) | 36/133 | 36/132 | 23/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy Treatment (N=133) | Adjunctive Treatment (N=132) | Laser Control (N=128)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0
Cataract (Fellow eye) (Eye disorders) | 1 | 2 | 0
Cataract (Study eye) (Eye disorders) | 0 | 2 | 0
Diabetic retinal oedema (Fellow eye) (Eye disorders) | 1 | 0 | 0
Diabetic retinopathy (Fellow eye) (Eye disorders) | 1 | 1 | 0
Maculopathy (Fellow eye) (Eye disorders) | 2 | 0 | 0
Retinal detachment (Fellow eye) (Eye disorders) | 0 | 1 | 0
Retinal detachment (Study eye) (Eye disorders) | 0 | 1 | 0
Retinal haemorrhage (Fellow eye) (Eye disorders) | 1 | 0 | 0
Vitreous haemorrhage (Fellow eye) (Eye disorders) | 2 | 0 | 1
Vitreous haemorrhage (Study eye) (Eye disorders) | 0 | 0 | 1
Epulis (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Polyp colorectal (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1
Conjunctivitis bacterial (Study eye) (Infections and infestations) | 0 | 1 | 0
Diabetic gangrene (Infections and infestations) | 0 | 0 | 1
Endophthalmitis (Study eye) (Infections and infestations) | 1 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Tuberculous pleurisy (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 2
Diabetic neuropathy (Study eye) (Nervous system disorders) | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy Treatment (N=133) | Adjunctive Treatment (N=132) | Laser Control (N=128)
Conjunctival haemorrhage (Study eye) (Eye disorders) | 17 | 12 | 7
Diabetic retinal oedema (Fellow eye) (Eye disorders) | 11 | 8 | 2
Nasopharyngitis (Infections and infestations) | 10 | 10 | 8
Hypertension (Vascular disorders) | 6 | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.